CLINICAL TRIAL: NCT01037673
Title: Does the Need of Arthroscopic Subacromial Decompression Change After Eccentric Physical Therapy Exercises in Patients With Subacromial Pain? - A Randomized Clinical Trial
Brief Title: Subacromial Impingement - The Need of Arthroscopic Subacromial Decompression After Eccentric Physical Therapy Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Kajsa Johansson, Senior lecturer, Linköping University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 88201401
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2009-12

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Resistance Training; Exercise; Exercise Movement Techniques; Posture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PT progressive exercises (Experimental): A progressive program of movement and strength exercises for the rotator cuff and scapular muscles combined with mobilisation of the joint capsule when needed
  Interventions: Procedure: Exercise program
- Movement exercises neck and shoulder (Active Comparator): General movements for the neck and shoulder,
  Interventions: Procedure: Exercise program; Procedure: Movement exercises

INTERVENTIONS:
Procedure: Exercise program — A progressive program where load and complexity increases during a 3 month period. Initially PT-tutored every week and then every other week.
  Other Names: Eccentric; Rotator cuff; Exercises; Scapular stabilization
Procedure: Movement exercises — A program with the same movements to maintain flexibility in the neck and shoulder. Initially PT-tutored every week and then every other week.
  Other Names: Exercises; posture
  Arms: Movement exercises neck and shoulder

SUMMARY:
Objective:

A randomized clinical trial in order to evaluate the efficacy of structured eccentric exercises tutored by a physical therapist (PT) for patients with subacromial impingement.

Hypothesis:

H1 The exercises has a satisfactory effect and the need of an arthroscopic subacromial decompression can be reconsidered.

H0 No difference between the two exercises (experimental and active control) and the patients still need surgery

Further the study objective is to evaluate predictors for a positive or negative treatment response after three months of rehabilitation as well as after 12 months.

Method:

Patients referred to the orthopedic unit for an arthroscopic subacromial decompression, are offered a three month rehabilitation program during the waiting time for surgery which is approximately 4-6 months. All patients must have tried conservative treatments for at least 6 months in primary care with unsatisfactory results. The patients will be randomized to either the structured eccentric exercises tutored by a physical therapist or control exercises with general movements for the neck and shoulders. All patients has an equal number of sessions with the PT to offer similar attention. After three months the following key-question has to be answered: due to your current experience of your shoulder problems do you still need this surgical intervention? A blinded orthopedic surgeon evaluates the following outcomes at baseline and after three and twelve months. Primary outcomes: Constant-Murley shoulder assessment, Disabilities of the Arm Shoulder and Hans and different aspects of pain. Secondary outcomes; EQ-5D, sick-leave and return to work. All patients are evaluated with a diagnostic ultrasound in order to reveal the condition of the rotator cuff. Also long-term results in those who go thorough with the surgery and those who decline will be assessed after 12 months.

Importance of the study results:

Since there is no consensus about which intervention that should be preferred for patients with subacromial impingement the results of the current study is warranted. If this exercise program is successful it can be implemented into clinical practice. Further, clinical characteristics of patients that really need an arthroscopic subacromial decompression can be identified.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial impingement verified with Neer impingement injection test
* At least 6 months duration
* Treated in primary care without satisfactory result for at least 6 months

Three of these five must be positive:

* Neer impingement sign
* Hawkins-Kennedy impingement sign
* Jobe supraspinatus test
* Patte maneuver
* Typical history and pain location (C5 dermatome)

Exclusion Criteria:

* Radiological finding of malignancy, osteoarthritis, fractures
* Polyarthritis or fibromyalgia
* Pathological hyper-laxity or dislocation of the any of the shoulder joints
* Cervical spine pathology
* Lack of communication skills that prevent the use of outcome measures

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Constant-Murley shoulder assessment | Baseline and change after three months of exercises, 3 month follow-up
  Measure a combination of self assessed and clinician assessed items; pain, range-of-motion (flexion and abduction), functional positions (hand in neck as well as hand in back), abduction strength.
  The score is summarized to a maximum of 100 for best available shoulder function.
Constant_Murley shoulder assessment | Change from baseline to the 12-month follow-up
  Measure a combination of self assessed and clinician assessed items; pain, range-of-motion (flexion and abduction), functional positions (hand in neck as well as hand in back), abduction strength.
  The score is summarized to a maximum of 100 for best available shoulder function.

SECONDARY OUTCOMES:
Health Related Quality of Life by EuroQol 5 dimensions | Baseline and change aftert three months of exercises
  Measures different items related to heath related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It results in a health-state where an index of 1 is optimal.
Health Related Quality of Life by EuroQol 5 dimensions | Change from baseline to the 12-month follow-up
  Measures different items related to heath related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It results in a health-state where an index of 1 is optimal.

CONTACTS AND LOCATIONS:
Overall Officials: Kajsa Johansson, PhD, RPT, Study Chair — Linkoeping University
Locations (1):
- University Hospital, Linköping, Sweden

REFERENCES:
- [Derived] Holmgren T, Hallgren HB, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. Br J Sports Med. 2014 Oct;48(19):1456-7. doi: 10.1136/bjsports-2014-e787rep. PMID 25213604
- [Derived] Hallgren HC, Holmgren T, Oberg B, Johansson K, Adolfsson LE. A specific exercise strategy reduced the need for surgery in subacromial pain patients. Br J Sports Med. 2014 Oct;48(19):1431-6. doi: 10.1136/bjsports-2013-093233. Epub 2014 Jun 26. PMID 24970843
- [Derived] Holmgren T, Bjornsson Hallgren H, Oberg B, Adolfsson L, Johansson K. Effect of specific exercise strategy on need for surgery in patients with subacromial impingement syndrome: randomised controlled study. BMJ. 2012 Feb 20;344:e787. doi: 10.1136/bmj.e787. PMID 22349588